CLINICAL TRIAL: NCT03996369
Title: A Phase 3, Randomized, Double-Blind, Placebo-Controlled, 12-Week Study to Assess the Efficacy and Safety of Etrasimod in Subjects With Moderately to Severely Active Ulcerative Colitis
Brief Title: Etrasimod Versus Placebo as Induction Therapy in Moderately to Severely Active Ulcerative Colitis
Acronym: ELEVATE UC 12
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Arena Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: APD334-302; 2018-003986-33 (EudraCT Number)
Record Dates: First submitted 2019-06-21; First posted 2019-06-24 (Actual); Results first posted 2022-12-21 (Actual); Last update posted 2022-12-21 (Actual); Status verified 2022-01

CONDITIONS: Ulcerative Colitis
Keywords: Ulcerative Colitis; Etrasimod; APD334
MeSH Terms: conditions — Colitis, Ulcerative | interventions — etrasimod

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Etrasimod 2 mg (Experimental)
  Interventions: Drug: Etrasimod
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Etrasimod — Etrasimod 2 mg tablet by mouth, once daily up to 12-Week Induction Treatment Period
  Other Names: APD334
  Arms: Etrasimod 2 mg
Drug: Placebo — Etrasimod matching placebo tablet by mouth, once daily up to 12-Week Induction Treatment Period
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the efficacy of etrasimod on clinical remission in participants with moderately to severely active ulcerative colitis (UC).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with ulcerative colitis (UC) ≥ 3 months prior to screening
* Active UC confirmed by endoscopy

Exclusion Criteria:

* Severe extensive colitis
* Diagnosis of Crohn's disease (CD) or indeterminate colitis or the presence or history of a fistula consistent with CD
* Diagnosis of microscopic colitis, ischemic colitis, or infectious colitis

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 354 (Actual)
Dates: Start 2020-09-15 (Actual); Primary Completion 2021-12-07 (Actual); Study Completion 2021-12-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arena CT.gov Administrator, Study Director — Arena Pharmaceuticals
Locations (406):
- United States (61):
  - Digestive Health Specialists of the Southeast, Dothan, Alabama
  - East View Medical Research, LLC, Mobile, Alabama
  - Arizona Digestive Health, Sun City, Arizona
  - Om Research, LLC, Lancaster, California
  - Entertainment Medical Group, Inc., Los Angeles, California
  - United Medical Doctors, Murrieta, California
  - ACRC Studies,LLC, San Diego, California
  - Paradigm Clinical Research Institute, Torrance, California
  - University of Colorado, Aurora, Colorado
  - Peak Gastroenterology Associates, Colorado Springs, Colorado
  - Gastro Florida, Clearwater, Florida
  - Florida Center for Gastroenterology, Largo, Florida
  - Global Life Research Network, LLC, Miami, Florida
  - Life Medical Center & Research, Inc, Miami Lakes, Florida
  - Gastroenterology Group of Naples, Naples, Florida
  - NSB Research, New Smyrna Beach, Florida
  - Pediatric & Adult Research Center, Orlando, Florida
  - IMIC, Inc., Palmetto Bay, Florida
  - Advanced Medical Research Center, Port Orange, Florida
  - Theia Clinical Research, LLC, St. Petersburg, Florida
  - Lenus Research & Medical Group, LLC, Sweetwater, Florida
  - USF Department of Surgery, Tampa, Florida
  - GCP Clinical Research, Tampa, Florida
  - Guardian Angel Research Center, Tampa, Florida
  - Florida Medical Clinic, P.A., Zephyrhills, Florida
  - Atlanta Gastroenterology Associates, Atlanta, Georgia
  - Children's Center for Digestive Health Care, LLC, Atlanta, Georgia
  - Atlanta Center for Gastroenterology, P.C., Decatur, Georgia
  - University of Chicago Medical Center, Chicago, Illinois
  - Illinois Gastroenterology Group, Gurnee, Illinois
  - Texas Digestive Disease Consultants, Baton Rouge, Louisiana
  - Chevy Chase Clinical Research, Chevy Chase, Maryland
  - Gastro Center of Maryland, Columbia, Maryland
  - West Michigan Clinical Research Center, Wyoming, Michigan
  - Washington University School of Medicine, St Louis, Missouri
  - Sierra Clinical Research, Las Vegas, Nevada
  - Las Vegas Medical Research, Las Vegas, Nevada
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Duke University Medical Center, Durham, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - Great Lakes Medical Research, LLC - Mentor, Mentor, Ohio
  - Care Access Research, Poland, Ohio
  - Great Lakes Medical Research, LLC - Harrisburg, Harrisburg, Pennsylvania
  - Tri-Cities Gastroenterology, Kingsport, Tennessee
  - GI for Kids, Knoxville, Tennessee
  - Texas Clinical Research Institute, LLC, Arlington, Texas
  - The University of Texas at Austin Dell Medical School, Austin, Texas
  - Texas Gastroenterology Associates, PA, Cypress, Texas
  - Texas Digestive Disease Consultants - Dallas, Dallas, Texas
  - DHAT Research Institute, Garland, Texas
  - Baylor Gastroenterology Assoc, Houston, Texas
  - Rio Grande Gastroenterology, McAllen, Texas
  - Texas Digestive Disease Consultants - San Marcos, San Marcos, Texas
  - Tyler Research Institute, LLC, Tyler, Texas
  - Victoria Gastroenterology, Victoria, Texas
  - Care Access Research LLC, Ogden, Utah
  - Blue Ridge Medical Research, Lynchburg, Virginia
  - Washington Gastroenterology, Bellevue, Washington
  - Virginia Mason, Seattle, Washington
  - Marshall University Department of Clinical Research, Huntington, West Virginia
  - Medical College of Wisconsin Clinical Trials Office, Milwaukee, Wisconsin
- Argentina (5):
  - Clinica Adventista Belgrano, CABA, Buenos Aires
  - Mautalen Salud e Investigacion, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - Fundación Respirar- Centro Médico Dra. De Salvo, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - Instituto de Investigaciones Clínicas Quilmes SRL, Quilmes, Buenos Aires
  - CICE Sanatorio 9 de Julio, San Miguel de Tucumán, Tucumán Province
- Australia (9):
  - Bankstown-Lidcombe Hospital, Bankstown, New South Wales
  - Nepean Hospital, Kingswood, New South Wales
  - Coastal Digestive Health, Maroochydore, Queensland
  - Coral Sea Clinical Research Institute, North Mackay, Queensland
  - Footscray Hospital, Footscray, Victoria
  - Austin Health, Heidelberg, Victoria
  - Royal Melbourne Hospital, Parkville, Victoria
  - Liverpool Hospital, Liverpool
  - Alfred Hospital, Melbourne
- Austria (3):
  - Lkh Univ. Klinikum Graz, Graz
  - KH der Barmherzigen Brüder Linz, Interne Abteilung, Linz
  - AKH - Medizinische Universität Wien, Vienna
- Belarus (4):
  - Grodno City Clinical Hospital #4, Grodno
  - Institution "Gomel Regional Clinical Hospital", Homyel
  - Vitebsk Regional Clinical Hospital, Vitebsk
  - Vitebsk Regional Clinical Specialized Center, Vitebsk
- Belgium (8):
  - University Hospital Antwerp Gastroenterology and Hepatology Department, Edegem, Antwerp
  - Dr. Peter Bossuyt - GI Clinical Research Center, Bonheiden
  - AZ Sint-Lucas & Volkskliniek, Ghent
  - UZ Gent - Gastroenterology, Ghent
  - UZ Leuven Campus Gasthuisberg, Leuven
  - AZ Sint-Maarten, Mechelen
  - ZNA Jan Palfijn, Merksem
  - AZ Delta, Roeselare
- Bulgaria (11):
  - UMHAT "Sv. Georgi", EAD, Plovdiv
  - UMHAT Kanev AD, Ruse, Rousse
  - Diagnostic-Consultative Center I - Sliven, EOOD, Sliven
  - ACIBADEM CITY CLINIC TOKUDA HOSPITAL EAD,Clinical Research Center, Sofia
  - DCC "Alexandrovska", EOOD, Sofia
  - UMHAT "Tsaritsa Yoanna-ISUL" EAD, Sofia
  - UMHATEM "N.I.Pirogov" EAD, Gastroenterology Department/Clinical Research center, Sofia
  - Diagnostic Consultation Center CONVEX EOOD, Sofia
  - Acibadem City Clinic University Hospital EOOD, Sofia
  - Medical center "Nov Rehabilitatsionen Tsentar" EOOD, Stara Zagora
  - Medical Centre MEDICA Plus OOD, Veliko Tarnovo
- Canada (2):
  - Heritage Medical Research Clinic, Calgary, Alberta
  - LHSC - University Hospital, London, Ontario
- Chile (5):
  - Enroll SpA, Santiago
  - Biomedica Research Group, Santiago
  - Hospital Sotero del Rio, Santiago
  - Centro de Investigación del Maule SPA, Talca
  - Clinical Research Chile SpA, Valdivia
- Colombia (4):
  - Clínica de la Costa Ltda., Barranquilla, Atlántico
  - Clinica de la Mujer Centro de Investigaciones, Bogota, Cundinamarca
  - Hospital San Juan de Dios Fundacion Cardiomet-Cequin, Armenia, Quindío Department
  - Clinica farallones centro de investigaciones clinicas CIC, Cali, Valle del Cauca Department
- Croatia (5):
  - General Hospital "Dr. Tomislav Bardek" Koprivnica, Koprivnica
  - Clinical Hospital Centre Osijek, Osijek
  - General Hospital Zadar, Zadar
  - Clinical Hospital Sveti Duh, Zagreb
  - University hospital centre Zagreb, Zagreb
- Czechia (10):
  - Fakultni nemocnice u svate Anny v Brne, Brno
  - Hepato Gastroenterologie HK s.r.o., Hradec Králové
  - GASTRO JeKa s.r.o., Klatovy
  - PreventaMed s.r.o., Olomouc
  - Fakultni nemocnice Ostrava, Ostrava-Poruba
  - Axon Clinical s. r. o., Prague
  - ISCARE I.V.F. a.s., Prague
  - Nemocnice Na Bulovce, Prague
  - Oblastni nemocnice Pribram a.s., Příbram
  - Nemocnice Slany, Slaný
- Denmark (2):
  - Aalborg University Hospital, department of medical gastroenterology, Aalborg, North Denmark
  - Herlev Hospital, Gastroenheden, 54Q2, Herlev
- Estonia (4):
  - Innomedica OÜ, Tallinn
  - West Tallinn Central Hospital, Tallinn
  - North Estonia Medical Centre Foundation, Tallinn
  - Tartu University Hospital, Tartu
- France (13):
  - CHU Nice - Hôpital de l'Archet 2, Nice, Alpes Maritimes
  - CHU Dijon - Hôpital Bocage Central, Dijon, Côte-d'Or
  - Hôpital Rangueil Service Gastro-entérologie et pancreatologie, Toulouse, Haute Garonne
  - CHU Montpellier - Hopital Saint Eloi, Montpellier, Herault
  - Chu Pontchaillou Rennes, Rennes, Ille Et Vilaine
  - CHU Nantes Hôtel-Dieu, Nantes, Loire Atlantique
  - CHRU-Nancy Brabois, Vandœuvre-lès-Nancy, Meurthe Et Moselle
  - CHU Lille - Hôpital Claude Huriez, Lille, Nord
  - CHU Clermont Ferrand - Hôpital d'Estaing, Clermont-Ferrand, Puy De Dome
  - Unite de Recherche Clinique-Urc, Montfermeil, Seine Saint Denis
  - Chu Amiens Picardie-Sit Sud, Amiens, Somme
  - Groupement Hospitalier Sud - Hôpital Bicêtre, Le Kremlin-Bicêtre, Val De Marne
  - CHU Grenoble Alpes - Hôpital Michallon, Grenoble
- Georgia (8):
  - LTD Acad. F. Todua Medical Centre, LTD. Research Institution of Clinical Medicine, Tbilisi
  - LTD Israeli-Georgian medical research clinic Helsicore, Tbilisi
  - LLC Vivamedi, Tbilisi
  - LTD Institute of Clinical Cardiology, Tbilisi
  - JSC Infectious Diseases, AIDS and Clinical Immunology Research Center, Tbilisi
  - LTD Aversi Clinic, Tbilisi
  - LTD Central University Clinic After Academic N. Kipshidze, Tbilisi
  - Malkhaz Katsiashvili Multiprofile Emergency Medicine Center, Tbilisi
- Germany (8):
  - Praxis Dr. Joergensen, Remscheid, North Rhine-Westphalia
  - Schwerpunktpraxis Bonn, Bonn, Rhineland-Palatinate
  - Clinic for Internal Medicine I, University hospital Schleswig-Holstein, Campus Kiel, Kiel, Schleswig-Holstein
  - Charité Universitätsmedizin Berlin - Campus Charité Mitte, Berlin
  - Krankenhaus Waldfriede, Berlin
  - Florence-Nightingale-Krankenhaus, Düsseldorf
  - Johanna Etienne Krankenhaus, Neuss
  - Klinische Forschung Schwerin GmbH, Schwerin
- Hungary (12):
  - DRC Gyogyszervizsgalo Kozpont Kft., Balatonfüred
  - Bekes Megyei Kozpont Korhaz Dr Rethy Pal Tagkorhaz, 4. Belgyogyaszat es 2. Gasztroenterologia, Békéscsaba
  - Obudai Egeszsegugyi Centrum Kft., Budapest
  - Endoexpert Egeszsegugyi Szolgaltato Kft, Budapest
  - Semmelweis Egyetem, II.sz. Belgyogyaszati Klinika, Budapest
  - Pannonia Maganorvosi Centrum, Budapest
  - Debreceni Egyetem Klinikai Kozpont Belgyogyaszati Klinika -Gasztroenterologia, Debrecen
  - Bugat Pal Korhaz, Gyöngyös
  - SZTE AOK I.st dept. of Internal Medicine., Szeged
  - Clinfan Ltd. Outpatient Clinic, Szekszárd
  - Dept of Gastroenterology, Szent Gyorgy Hospital, Székesfehérvár
  - Szent Borbala Korhaz, Tatabánya
- India (10):
  - Nirmal Hospitals Pvt Ltd, Surat, Gujarat
  - Surat Institute of Digestive Sciences, Surat, Gujarat
  - Fortis Memorial Research Institute, Gurgaon, Haryana
  - All India Institute of Medical Sciences, Kochi, Kerala
  - Aster Medcity,Aster DM healthcare Ltd, Kochi, Kerala
  - Government Medical College and Super Speciality Hospital, Nagpur, Maharashtra
  - Midas Multispeciality Hospital Pvt.Ltd., Nagpur, Maharashtra
  - Ruby Hall Clinic, Pune, Maharashtra
  - Shweta Paliwal/Vipin Kumar Jain, Jaipur, Rajasthan
  - Postgraduate department of Medicine, GSVM Medical college, Kanpur, Uttar Pradesh
- Israel (9):
  - HaEmek Medical Center, Afula
  - Bnei Zion Medical Center, Haifa
  - Wolfson Medical Center, Holon
  - Shaare Zedek Medical Center, Jerusalem
  - Hadassah University Hospital - Ein Kerem, Jerusalem
  - Galilee Medical Center, Nahariya
  - Rabin Medical Center-Beilinson Campus, Petah Tikva
  - Chaim Sheba Medical Center, Ramat Gan
  - Kaplan Medical Center, Rehovot
- Italy (16):
  - Azienda Ospedaliera Saverio De Bellis, Castellana Grotte, Bari
  - Ospedale di Circolo, Rho, Milano
  - Istituto Clinico Humanitas, Rozzano, Milano
  - I.R.C.C.S Policlinico San Donato, San Donato Milanese, Milano
  - Ospedale Sacro Cuore Don Calabria, Negrar, Verona
  - Azienda Ospedaliera Universitaria Policlinico Sant'Orsola Malpighi, Bologna
  - Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia (Presidio Spedali Civili), Brescia
  - Azienda Ospedaliera Ospedale Cannizzaro, Catania
  - Azienda Ospedaliero Universitaria Mater Domini, Catanzaro
  - Azienda Ospedaliera Universitaria Careggi, Florence
  - A.O.U. Policlinico di Modena, Modena
  - Ospedale Sandro Pertini, Roma
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS - CEMAD, Roma
  - A.O. Ordine Mauriziano di Torino - P.O. Ospedale Umberto I, Torino
  - Centro Ricerche Cliniche di Verona, Verona
  - Ospedale San Bortolo di Vicenza, Vicenza
- Japan (60):
  - Koujunkai Daido Clinic, Nagoya, Aichi-ken
  - Nagoya City University Hospital, Nagoya, Aichi-ken
  - Toyohashi Municipal Hospital, Toyohashi, Aichi-ken
  - NHO Hirosaki National Hospital, Hirosaki-shi, Aomori
  - Hirosaki University Hospital, Hirosaki-shi, Aomori
  - Tsujinaka Hospital Kashiwanoha, Kashiwa, Chiba
  - Saiseikai Matsuyama Hospital, Matsuyama, Ehime
  - Ehime University Hospital, Toon-shi, Ehime
  - Fukuoka Tokushukai Hospital, Kasuga, Fukuoka
  - JCHO Kyushu Hospital, Kitakyushu-shi, Fukuoka
  - Kurume University Hospital, Kurume-shi, Fukuoka
  - Fukushima Medical University Hospital, Fukushima, Fukushima
  - Gifu University Hospital, Gifu, Gifu
  - Ogaki Municipal Hospital, Ogaki-shi, Gifu
  - SUBARU Health Insurance Society Ota Memorial Hospital, Ota-shi, Gunma
  - NHO Fukuyama Medical Center, Fukuyama-shi, Hiroshima
  - Hiroshima City Hiroshima Citizens Hospital, Hiroshima, Hiroshima
  - Hiroshima University Hospital, Hiroshima, Hiroshima
  - Asahikawa City Hospital, Asahikawa-shi, Hokkaido
  - Tokushukai Sapporo Tokushukai Hospital, Sapporo, Hokkaido
  - Sapporo-Kosei General Hospital, Sapporo, Hokkaido
  - NHO Mito Medical Center, Higashi, Ibaraki
  - Yuai Memorial Hospital, Koga-shi, Ibaraki
  - Tsuchiura Kyodo General Hospital, Tsuchiura-shi, Ibaraki
  - NHO Kanazawa Medical Center, Kanazawa, Ishikawa-ken
  - Iwate Medical University Uchimaru Medical Center, Morioka, Iwate
  - Takamatsu Red Cross Hospital, Takamatsu, Kagawa-ken
  - Kagawa Prefectural Central Hospital, Takamatsu, Kagawa-ken
  - Jiaikai Izuro Imamura Hospital, Kagoshima, Kagoshima-ken
  - Sameshima Hospital, Kagoshima, Kagoshima-ken
  - Gokeikai Ofuna Chuo Hospital, Kamakura-shi, Kanagawa
  - Sagamihara Kyodo Hospital, Sagamihara-shi, Kanagawa
  - NHO Yokohama Medical Center, Yokohama, Kanagawa
  - Japanese Red Cross Kumamoto Hospital, Kumamoto, Kumamoto
  - NHO Kyoto Medical Center, Kyoto, Kyoto
  - Mie University Hospital, Tsu, Mie-ken
  - Mie Prefectural General Medical Center, Yokkaichi, Mie-ken
  - Tohoku University Hospital, Sendai, Miyagi
  - JOHAS Tohoku Rosai Hospital, Sendai, Miyagi
  - Sendai City Hospital, Sendai, Miyagi
  - Nara Medical University Hospital, Kashihara, Nara
  - Saiseikai Niigata Hospital, Niigata, Niigata
  - Kansai Medical University Hospital, Hirakata-shi, Osaka
  - Tokushukai Kishiwada Tokushukai Hospital, Kishiwada-shi, Osaka
  - Osaka City University Hospital, Osaka, Osaka
  - Japan Community Health care Organization Osaka Hospital, Osaka, Osaka
  - Osaka Medical College Hospital, Takatsuki-shi, Osaka
  - Saga University Hospital, Saga, Saga-ken
  - JCHO Saitama Medical Center, Saitama-shi, Saitama
  - Shiga University of Medical Science Hospital, Ōtsu, Shiga
  - St. Luke's International Hospital, Chuo -ku, Tokyo
  - Teikyo University Hospital, Itabashi-ku, Tokyo
  - Showa General Hospital, Kodaira-shi, Tokyo
  - Jikei University Hospital, Minato-ku, Tokyo
  - Kitasato University Kitasato Institute Hospital, Minato-ku, Tokyo
  - NTT Medical Center Tokyo, Shinagawa-ku, Tokyo
  - JCHO Tokyo Yamate Medical Center, Shinjuku-ku, Tokyo
  - Toyama Prefectural Central Hospital, Toyama, Toyama
  - Wakayama Medical University Hospital, Wakayama, Wakayama
  - Fukuoka University Hospital, Fukuoka
- Lebanon (3):
  - Saint George Hospital University Medical Center, Beirut
  - American University of Beirut Medical Center, Beirut
  - Hotel Dieu de France Hospital, Beirut
- Lithuania (3):
  - Republican Panevezys Hospital, Department of Gastroenterology, Panevezys
  - UAB "Inlita", Santaros Clinical Trials Centre, Vilnius
  - Vilnius University Hospital Santaros Clinics, Center of Hepatology, Gastroenterology and Dietology, Vilnius
- Mexico (6):
  - Consultorio Medico, InvesclinicMX, Irapuato, Guanajuato
  - Centro de Investigacion Medico Biologica y Terapia Avanzada s.c., Guadalajara, Jalisco
  - InspirePharma S. de R. L. de C.V., Monterrey, Nuevo León
  - Scientia Investigación Clínica S.C., Chihuahua City
  - Hospital Angeles Chihuahua, Chihuahua City
  - Faicic S. de R.L. de Cv, Veracruz
- Moldova (4):
  - Republican Clinical Hospital, ARENSIA Exploratory Medicine, Chisinau
  - Rtl Sm Srl, Chisinau
  - Timofei Mosneaga Republican Clinical Hospital, Department of Gastroenterology, Chisinau
  - RTL SM SRL, Institutia Medico- Sanitara Publica Spitalul Clinic, Sectia Proctologie, Chisinau
- Netherlands (3):
  - Zuyderland Medisch Centrum - Sittard-Geleen, Geleen
  - Radboudumc, Nijmegen
  - ETZ Elisabeth, Tilburg
- Poland (21):
  - Centrum Dentystyczno-Lekarskie Promedica Joanna Markiewicz, Będzin
  - Gastromed Kralisz, Romatowski, Stachurska sp.j, Bialystok
  - Centrum Medyczne Pratia Czestochowa, Częstochowa
  - Karkonoskie Centrum Badan Klinicznych Lexmedica, Jelenia Góra
  - Centrum Medyczne Plejady, Krakow
  - Topolowa Medicenter Mrozek & Wspolnicy Spolka Jawna, Krakow
  - AmiCare Sp. z O.O. Sp.K., Lodz
  - IP Clinic, Lodz
  - Allmedica Badania Kliniczne Sp. z o.o. Sp.k., Nowy Targ
  - Medicome Sp. Zo.O., Oświęcim
  - Centrum Medyczne Grunwald, Poznan
  - SOLUMED Centrum Medyczne, Poznan
  - Korczowski Bartosz, Gabinet Lekarski, Rzeszów
  - Centrum Medyczne Medyk, Rzeszów
  - ENDOSKOPIA Sp.zo.o, Sopot
  - DC-MED, Swidnica
  - Twoja Przychodnia-Szczecinskie Centrum Medyczne, Szczecin
  - Centrum Zdrowia MDM, Warsaw
  - Centralny Szpital Kliniczny MSW w Warszawie, Warsaw
  - EMC INSTYTUT MEDYCZNY SA, EuroMediCare Szpital Specjalistyczny z Przychodnia - Dzial Farmacji, Wroclaw
  - Centrum Medyczne Oporow, Wroclaw
- Portugal (6):
  - Hospital de Braga, Braga
  - Centro Hospitalar e Universitário de Coimbra Serviço Gastrenterologia, Coimbra
  - Hospital da Senhora da Oliveira Guimarães, Guimarães
  - Hospital da Luz Lisboa, Lisbon
  - Centro Hospitalar de São João, EPE, Porto
  - Centro Hospitalar de Vila Nova de Gaia/Espinho, E.P.E, Vila Nova de Gaia
- Romania (10):
  - S.C MedLife SA, Bucharest
  - S.C Delta Health Care S.R.L, Ponderas Academic Hospital, Bucharest
  - S.C Euroclinic Hospital S.A, Bucharest
  - Spitalul Clinic Colentina, Bucharest
  - Institutul Clinic Fundeni, Bucharest
  - S.C Policlinica CCBR S.R.L, Bucharest
  - S.C. Centrul Medical Unirea SRL, Bucharest
  - Spitalul Clinic Judetean de Urgenta Cluj Napoca, Cluj-Napoca
  - Spitalul Clinic Judetean de Urgenta Craiova, Craiova
  - S.C Pelican Impex S.R.L, Oradea
- Russia (20):
  - LLC "Multidisciplinary Medical Clinic "Anthurium", Barnaul
  - LLC "Alyans Biomedical- Ural Group", Izhevsk
  - Kazan State Medical University, Kazan'
  - SAIH "Kemerovo Regional Clinical Hospital", Kemerovo
  - SBIH of Nizhniy Novgorod region "Nizhniy Novgorod Regional Clinical Hospital n.a. N.A. Semashko", Nizhny Novgorod
  - LLC Medicine Center SibNovoMed, Novosibirsk
  - CDC "Ultramed", Omsk
  - State Budgetary Healthcare Institution "Penza Region Clinical Hospital n.a. N.N. Burdenko", Penza
  - Federal state Budgetary Educational Institution of Higher Education "North-Western Medical University", Saint Petersburg
  - FSBI of higher Education "First Saint Petersburg State Medical University n.a. I.P.Pavlov, Saint Petersburg
  - LLC "Gastroenterological centre Expert", Saint Petersburg
  - LLC SM-Clinic, Saint-Peterburg
  - Irkutsk State Medical Academy of Continuing Education, Samara
  - Private Educational Institution of Higher Education "Medical University "REAVIZ", Samara
  - LLC Medical Company "Hepatologist", Samara
  - SPb SBIH "City Hospital # 40 of Kurortnyi region", Sestroretsk
  - LLC Uromed, Smolensk
  - Stavropol Regional Clinical Diagnostic Centre, Stavropol
  - LLC "Polyclinic of ultrasonography 4D", Stavropol
  - City Clinical Hospital #8, Yaroslavl
- Serbia (6):
  - Clinical Center " Dr Dragisa Misovic Dedinje", Belgrade
  - Clinical Center of Serbia, Belgrade
  - Clinical Health Center Zvezdara, Belgrade
  - Clinical Center Bezanijska Kosa, Belgrade
  - Clinical Center Kragujevac, Kragujevac
  - General Hospital Sremska Mitrovica, Sremska Mitrovica
- Slovakia (8):
  - Endomed, S.R.O, Vranov nad Topľou, Presov
  - Fakultna nemocnica s poliklinikou F.D. Roosevelta, Banská Bystrica
  - Alian S.R.O, Bardejov
  - KM Management spol. s r.o., Nitra
  - Fakultna nemocnica Nitra, Nitra
  - Gastro I, s.r.o., Prešov
  - Accout Center s.r.o., Šahy
  - BeneDig s.r.o., Žilina
- South Africa (4):
  - Johese Clinical Research: Unitas, Lyttelton, Centurion
  - Johese Clinical Research, Midstream, Centurion
  - Lenasia Clinical Trial Centre, Lenasia, Gauteng
  - Dr JP Wright Practice, Cape Town, Western Cape
- South Korea (6):
  - Kyungpook National University Hospital, Junggu, Daegu
  - Yonsei University Wonju Severance Christian Hospital, Wŏnju, Gangwon-do
  - The Catholic University of Korea St. Vincent's Hospital, Suwon, Gyeonggi-do
  - Severance Hospital, Yonsei University Health System, Seoul, Seodaemun-gu
  - Dong-A University Hospital, Busan
  - Kyungpook National University Chilgok Hospital, Daegu
- Spain (5):
  - Hospital General Universitario de Alicante, Alicante
  - Centro Médico Teknon, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Universitario de Gran Canaria Dr. Negrin, Las Palmas
  - Hospital Universitario La Paz, Madrid
- Switzerland (3):
  - Kantonsspital Baden, Baden
  - Inselspital, Gaby Saner, Gastroenterologie, Bauchzentrum, Bern
  - Berner IBD study group c/o Gastroenterologische Praxis Balsiger, Seibold &Partner, Bern
- Thailand (3):
  - Siriraj Hospital, Bangkoknoi, Bangkok
  - King Chulalongkorn Memorial Hospital, Pathum Wan, Bangkok
  - Phramongkutklao Hospital, Ratchathewi, Bangkok
- Turkey (Türkiye) (6):
  - Uludag University Medical Faculty, Beşevler, Yenimahalle/Ankara
  - Hacettepe University Medical Faculty, Ankara
  - Gazi University Medical Faculty, Ankara
  - Antalya Training and Research Hospital, Antalya
  - Kocaeli University Research and Training Hospital, Kocaeli
  - Karadeniz Tecnical Uni. Med. Fac., Trabzon
- Ukraine (16):
  - I.I.Mechnykov Dnipropetrovsk Regional Clinical Hospital, Dnipro
  - Department of Propaedeutics of Internal Medicine Ivano-Frankivsk National Medical University, Ivano-Frankivsk
  - Municipal non-profit enterprise Regional Clinical Hospital of Ivano-Frankivsk Regional Council, Ga, Ivano-Frankivsk
  - CNE Prof. O.O. Shalimov Kharkiv City Clinical Hospital #2 of KCC, Kharkiv
  - Communal Non-commercial Enterprise of Kharkiv Regional Council Regional Clinical Hospital, Kharkiv
  - Communal Non-Commercial Enterprise City Clinical Hospital #13 of Kharkiv City Council, Kharkiv
  - Communal Noncommercial Enterprise Ye.Ye. Karabelesh Kherson City Clinical Hospital of Kherson City, Kherson
  - Kremenchuk first city hospital n.a. O.T. Bohaievskyi, Kremenchuk
  - Kyiv CCH #18 Dept of Proctology O. O. Bogomolets NMU, Kyiv
  - Kyiv City Clinical Hospital N 1, Kyiv
  - Communal Non-Commercial Enterprise Lviv Clinical Hospital of Emergency Medical Care, Lviv
  - Odesa regional clinical hospital, regional center of gastroenterology, surgical department, Odesa
  - A. Novak Transcarpathian Regional Clinical Hospital, Uzhhorod
  - Medical Clinical Investigational Center of Medical Center Health Clinic LLC, Vinnytsia
  - M.I. Pyrogov VRCH Dept of Gastroenterology M.I. Pyrogov VNMU, Vinnytsia
  - SRI of Invalid Rehabilitation (EST Complex) of Vinnytsia M.I.Pyrogov NMU MOHU, Vinnytsia
- United Kingdom (4):
  - Whipps Cross University Hospital, London, Greater London
  - Guy's and Saint Thomas NHS Foundation Trust, London, Greater London
  - Norfolk and Norwich University Hospital, Norwich, Norfolk
  - Yeovil District Hospital, Yeovil, Somerset

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dubinsky MC, Chaparro M, Irving PM, Hur P, Sidhu S, Woolcott JC, Wang W, Goetsch M, Torres J, Panaccione R. Rapid symptomatic improvement with etrasimod in ulcerative colitis: a post-hoc analysis of the ELEVATE UC program. Inflamm Bowel Dis. 2026 Feb 8:izaf333. doi: 10.1093/ibd/izaf333. Online ahead of print. PMID 41655066
- [Derived] Chaparro M, Panaccione R, Sands BE, Irving PM, Goetsch M, Kunina E, Wang W, Wu J, Woolcott JC, Bartolome L, Cognata C, Wosik K, Dubinsky MC. Etrasimod for the symptomatic relief of ulcerative colitis: a post-hoc analysis from the ELEVATE UC clinical programme. BMJ Open Gastroenterol. 2025 Aug 31;12(1):e001838. doi: 10.1136/bmjgast-2025-001838. PMID 40889900
- [Derived] Yarur AJ, Reinisch W, Chang S, Gecse KB, Green J, Abbatemarco AM, Wu J, Goetsch M, Lazin K, Pradeep G, Sands BE. Efficacy of Etrasimod in Ulcerative Colitis: Analysis of ELEVATE UC 52 and ELEVATE UC 12 by Baseline Endoscopic Severity. Clin Gastroenterol Hepatol. 2026 Jan;24(1):210-220.e3. doi: 10.1016/j.cgh.2025.06.020. Epub 2025 Jul 4. PMID 40618942
- [Derived] Lichtenstein GR, Allegretti JR, Loftus EV Jr, Irving PM, Banerjee R, Charabaty A, Kuehbacher T, Bananis E, Woolcott JC, Dalam AB, Lazin K, Keating M, McDonnell A, Danese S. Assessment and Impact of Age on the Safety and Efficacy of Etrasimod in Patients With Ulcerative Colitis: A Post Hoc Analysis of Data From the ELEVATE UC Clinical Program. Inflamm Bowel Dis. 2025 Sep 1;31(9):2352-2362. doi: 10.1093/ibd/izae308. PMID 40184206
- [Derived] Sands BE, Dubinsky MC, Kotze PG, Vermeire S, Panaccione R, Long MD, Woolcott JC, Wu J, McDonnell A, Goetsch M, Bananis E, Yarur AJ. Efficacy and Safety of Etrasimod in Patients With Moderately to Severely Active Ulcerative Colitis Stratified by Baseline Modified Mayo Score: A Post Hoc Analysis From the Phase 3 ELEVATE UC Clinical Program. Inflamm Bowel Dis. 2025 Oct 1;31(10):2681-2692. doi: 10.1093/ibd/izaf036. PMID 40036804
- [Derived] Afzali A, Regueiro M, Yarur AJ, Zabana Y, Ng SC, Menon S, McDonnell A, Lazin K, Keating M, Bhattacharjee A, Branquinho D, Bananis E, Peyrin-Biroulet L. Concomitant Use of Etrasimod With Opioids or Antidepressants in Patients With Ulcerative Colitis-A Safety Analysis. United European Gastroenterol J. 2025 Jun;13(5):719-727. doi: 10.1002/ueg2.12745. Epub 2025 Feb 1. PMID 39891572
- [Derived] Yarur AJ, Long MD, Torres J, Nandi N, Cross RK, Abbatemarco AM, Blanco D, Niezychowski W, Crosby C, Wu J, Pradeep G, Goetsch M, Panaccione R. Body Mass Index Did Not Affect Efficacy and Safety of Etrasimod: A Post Hoc Analysis of the ELEVATE Ulcerative Colitis Clinical Program. Am J Gastroenterol. 2025 Nov 1;120(11):2611-2622. doi: 10.14309/ajg.0000000000003330. Epub 2025 Jan 29. PMID 39878434
- [Derived] Vermeire S, Rubin DT, Peyrin-Biroulet L, Dubinsky MC, Regueiro M, Irving PM, Goetsch M, Lazin K, Gu G, Wu J, Modesto I, McDonnell A, Guo X, Green J, Dalam AB, Yarur AJ. Cardiovascular events observed among patients in the etrasimod clinical programme: an integrated safety analysis of patients with moderately to severely active ulcerative colitis. BMJ Open Gastroenterol. 2025 Jan 8;12(1):e001516. doi: 10.1136/bmjgast-2024-001516. PMID 39778975
- [Derived] Yarur AJ, Chiorean MV, Allegretti JR, Cross RK, Ha C, Goetsch M, McDonnell A, Dalam AB, Wu J, Blanco DA, Abbatemarco AM, Panes J. Etrasimod as a Monotherapy or With Concomitant Use of Corticosteroids and/or Aminosalicylates: Results From the ELEVATE UC Clinical Program. Inflamm Bowel Dis. 2025 Aug 1;31(8):2144-2153. doi: 10.1093/ibd/izae288. PMID 39671695
- [Derived] Lees CW, Torres J, Leung Y, Vermeire S, Fellmann M, Modesto I, McDonnell A, Lazin K, Keating M, Goetsch M, Wu J, Loftus EV Jr. Non-serious adverse events in patients with ulcerative colitis receiving etrasimod: an analysis of the phase II OASIS and phase III ELEVATE UC 52 and ELEVATE UC 12 clinical trials. Therap Adv Gastroenterol. 2024 Nov 7;17:17562848241293643. doi: 10.1177/17562848241293643. eCollection 2024. PMID 39526078
- [Derived] Armuzzi A, Rubin DT, Schreiber S, Panes J, Fellmann M, Bartolome L, Gruben D, Goetsch M, Bhattacharjee A, Chaparro M, Dubinsky MC. Health-Related Quality of Life Outcomes With Etrasimod Treatment in Patients With Ulcerative Colitis: A Post Hoc Analysis of Data From ELEVATE UC 52 and ELEVATE UC 12. Inflamm Bowel Dis. 2025 Jun 13;31(6):1583-1594. doi: 10.1093/ibd/izae229. PMID 39326009
- [Derived] Sands BE, Leung Y, Rubin DT, Gecse KB, Panes J, Goetsch M, Wang W, Woolcott JC, Smith CC, Wosik K, Schreiber S. Etrasimod Corticosteroid-Free Efficacy, Impact of Concomitant Corticosteroids on Efficacy and Safety, and Corticosteroid-Sparing Effect in Ulcerative Colitis: Analyses of the ELEVATE UC Clinical Program. J Crohns Colitis. 2025 Mar 5;19(3):jjae150. doi: 10.1093/ecco-jcc/jjae150. PMID 39306680
- [Derived] Magro F, Peyrin-Biroulet L, Sands BE, Danese S, Jairath V, Goetsch M, Bhattacharjee A, Wu J, Branquinho D, Modesto I, Feagan BG. Endoscopic, Histologic, and Composite Endpoints in Patients With Ulcerative Colitis Treated With Etrasimod. Clin Gastroenterol Hepatol. 2025 Feb;23(2):341-350.e6. doi: 10.1016/j.cgh.2024.07.010. Epub 2024 Jul 31. PMID 39089519
- [Derived] Vermeire S, Sands BE, Peyrin-Biroulet L, D'Haens GR, Panes J, Yarur AJ, Wolf DC, Ritter T, Schreiber S, Woolcott JC, Modesto I, Keating M, Shan K, Wu J, Chiorean MV, Baert F, Dubinsky MC, Goetsch M, Danese S, Feagan BG. Impact of Prior Biologic or Janus Kinase Inhibitor Therapy on Efficacy and Safety of Etrasimod in the ELEVATE UC 52 and ELEVATE UC 12 Trials. J Crohns Colitis. 2024 Nov 4;18(11):1780-1794. doi: 10.1093/ecco-jcc/jjae079. PMID 38877972
- [Derived] Regueiro M, Siegmund B, Yarur AJ, Steinwurz F, Gecse KB, Goetsch M, Bhattacharjee A, Wu J, Green J, McDonnell A, Crosby C, Lazin K, Branquinho D, Modesto I, Abreu MT. Etrasimod for the Treatment of Ulcerative Colitis: Analysis of Infection Events from the ELEVATE UC Clinical Programme. J Crohns Colitis. 2024 Oct 15;18(10):1596-1605. doi: 10.1093/ecco-jcc/jjae060. PMID 38700040
- [Derived] Peyrin-Biroulet L, Dubinsky MC, Sands BE, Panes J, Schreiber S, Reinisch W, Feagan BG, Danese S, Yarur AJ, D'Haens GR, Goetsch M, Wosik K, Keating M, Lazin K, Wu J, Modesto I, McDonnell A, Bartolome L, Vermeire S. Efficacy and Safety of Etrasimod in Patients with Moderately to Severely Active Isolated Proctitis: Results From the Phase 3 ELEVATE UC Clinical Programme. J Crohns Colitis. 2024 Aug 14;18(8):1270-1282. doi: 10.1093/ecco-jcc/jjae038. PMID 38613425
- [Derived] Sandborn WJ, Vermeire S, Peyrin-Biroulet L, Dubinsky MC, Panes J, Yarur A, Ritter T, Baert F, Schreiber S, Sloan S, Cataldi F, Shan K, Rabbat CJ, Chiorean M, Wolf DC, Sands BE, D'Haens G, Danese S, Goetsch M, Feagan BG. Etrasimod as induction and maintenance therapy for ulcerative colitis (ELEVATE): two randomised, double-blind, placebo-controlled, phase 3 studies. Lancet. 2023 Apr 8;401(10383):1159-1171. doi: 10.1016/S0140-6736(23)00061-2. Epub 2023 Mar 2. PMID 36871574

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study included a screening period (up to 28 days), a double-blind induction treatment period (12 weeks), and a 2-week and a 4-week follow-up period. The target population consisted of male or female participants aged between 16 and 80 years (inclusive), with moderately to severely active ulcerative colitis (UC).
Pre-assignment Details: During the screening period, participants were evaluated for study entry based on the inclusion and exclusion criteria. Screening procedures to evaluate participant eligibility for the study were to be conducted within 28 days prior to study intervention administration on Day 1.
Groups:
- Etrasimod 2 mg: Participants were administered one tablet of etrasimod 2 milligrams (mg) orally once daily (QD) for 12 weeks.
- Placebo: Participants were administered one tablet of placebo orally QD for 12 weeks.
Period: Overall Study
Arm/Group | Etrasimod 2 mg | Placebo
Started | 238 | 116
Completed | 213 | 103
Not Completed | 25 | 13
Not completed — Protocol deviation | 1 | 1
Not completed — Physician Decision | 4 | 2
Not completed — Participant decision | 0 | 1
Not completed — Lack of Efficacy | 4 | 0
Not completed — Adverse Event | 9 | 0
Not completed — Withdrawal by Subject | 6 | 8
Not completed — Didn't meet Inclusion/Exclusion criteria | 1 | 0
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Population: Full Analysis Set: All randomized participants who received at least 1 dose of study intervention.
Groups:
- Total: Total of all reporting groups
Arm/Group | Etrasimod 2 mg | Placebo | Total
Number analyzed (Participants) | 238 | 116 | 354
Age, Continuous [Mean (Standard Deviation); unit: Years] | 40.3 (13.49) | 40.4 (13.28) | 40.4 (13.40)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 103 | 43 | 146
  Male | 135 | 73 | 208
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 9 | 19
  Not Hispanic or Latino | 226 | 107 | 333
  Unknown or Not Reported | 2 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 6 | 1 | 7
  Asian | 47 | 25 | 72
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 2 | 4
  White | 176 | 88 | 264
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 6 | 0 | 6

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Clinical Remission
Description: Clinical remission was based on the modified Mayo score (MMS). The MMS is a composite score of 3 assessments consisting of participant-reported symptoms using daily electronic (e)-diary and centrally read endoscopy: stool frequency (SF), rectal bleeding (RB) and endoscopic score (ES). Clinical remission was defined as SF sub-score = 0 (or = 1 with a greater than or equal to [>=] 1-point decrease from Baseline), RB sub-score = 0, and ES less than or equal to (<=) 1 (excluding friability). Each component sub-score ranged from 0 to 3 and total score range of the MMS was from 0 to 9, with higher scores indicating more severe disease.
Time Frame: Week 12
Population: Full Analysis Set Population (All randomized participants who received at least 1 dose of study intervention), with actual Baseline MMS 5 to 9. Only those participants with data available at the specified time points were analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | Etrasimod 2 mg | Placebo
Number analyzed (Participants) | 222 | 112
Percentage of participants | 24.8 | 15.2
Statistical Analysis 1: Comparison: Etrasimod 2 mg vs Placebo; Week 12; Test type: Superiority; p = 0.026, Cochran-Mantel-Haenszel; Risk Difference (RD) = 9.69, 95% CI 2-sided [1.14 to 18.23]

2. Secondary Outcome: Percentage of Participants Achieving Endoscopic Improvement
Description: Endoscopic improvement was defined as an ES <= 1 (excluding friability). The ES ranged from 0 to 3 (where 0 = normal/inactive disease and 3 = severe disease); higher score indicated more severe disease.
Time Frame: Week 12
Population: Full Analysis Set Population with actual Baseline MMS 5 to 9. Only those participants with data available at the specified time points were analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | Etrasimod 2 mg | Placebo
Number analyzed (Participants) | 222 | 112
Percentage of participants | 30.6 | 18.8
Statistical Analysis 1: Comparison: Etrasimod 2 mg vs Placebo; Week 12; Test type: Superiority; p = 0.009, Cochran-Mantel-Haenszel; Risk Difference (RD) = 12.11, 95% CI 2-sided [3.00 to 21.23]

3. Secondary Outcome: Percentage of Participants Achieving Symptomatic Remission
Description: Symptomatic remission was defined as an SF sub-score = 0 (or = 1 with a >= 1 point decrease from Baseline) and RB sub-score = 0. The SF sub-score ranged from 0 to 3 (where 0 = normal number of stools and 3 = at least 5 stools more than normal) and RB sub-score ranged from 0 to 3 (where 0 = no blood and 3 = blood alone passes). Higher scores indicated more severe disease.
Time Frame: Week 12
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Etrasimod 2 mg | Placebo
Number analyzed (Participants) | 222 | 112
Percentage of participants | 46.8 | 29.5
Statistical Analysis 1: Comparison: Etrasimod 2 mg vs Placebo; Week 12; Test type: Superiority; p = 0.001, Cochran-Mantel-Haenszel; Risk Difference (RD) = 17.48, 95% CI 2-sided [6.81 to 28.15]

4. Secondary Outcome: Percentage of Participants With Mucosal Healing
Description: Mucosal healing was defined as an ES <= 1 (excluding friability) with histologic remission measured by a Geboes Index score less than [<] 2.0). The ES ranged from 0 to 3 (where 0 = normal/inactive disease and 3 = severe disease). The Geboes score grading system, was a validated score for evaluating histologic disease activity in UC as follows: grade 0 = structural and architectural changes; grade 1 = chronic inflammatory infiltrate; grade 2 = lamina propria neutrophils and eosinophils; grade 3 = neutrophils in the epithelium; grade 4 = crypt destruction; grade 5 = erosions or ulceration. A higher Geboes score indicated more severe disease.
Time Frame: Week 12
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Etrasimod 2 mg | Placebo
Number analyzed (Participants) | 222 | 112
Percentage of participants | 16.2 | 8.9
Statistical Analysis 1: Comparison: Etrasimod 2 mg vs Placebo; Week 12; Test type: Superiority; p = 0.036, Cochran-Mantel-Haenszel; Risk Difference (RD) = 7.44, 95% CI 2-sided [0.50 to 14.39]

5. Secondary Outcome: Percentage of Participants Achieving Clinical Response
Description: Clinical response was based on the MMS which is a composite score of 3 assessments: SF, RB and ES. Clinical response was defined as a >= 2-point and >= 30 percent (%) decrease from Baseline MMS, and a >= 1-point decrease from Baseline in RB sub-score or an absolute RB sub-score <= 1. Each component sub-score ranged from 0 to 3 and total score range of the MMS was from 0 to 9, with higher scores indicating more severe disease.
Time Frame: Week 12
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Etrasimod 2 mg | Placebo
Number analyzed (Participants) | 222 | 112
Percentage of participants | 62.2 | 41.1
Statistical Analysis 1: Comparison: Etrasimod 2 mg vs Placebo; Week 12; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Risk Difference (RD) = 21.23, 95% CI 2-sided [10.18 to 32.29]

6. Secondary Outcome: Percentage of Participants Achieving Endoscopic Normalization
Description: Endoscopic normalization was defined as an ES = 0. The ES ranged from 0 to 3 (where 0= normal/inactive disease and 3= severe disease); higher score indicated more severe disease.
Time Frame: Week 12
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Etrasimod 2 mg | Placebo
Number analyzed (Participants) | 222 | 112
Percentage of participants | 17.1 | 8.0
Statistical Analysis 1: Comparison: Etrasimod 2 mg vs Placebo; Week 12; Test type: Superiority; p = 0.009, Cochran-Mantel-Haenszel; Risk Difference (RD) = 9.24, 95% CI 2-sided [2.27 to 16.20]

7. Secondary Outcome: Percentage of Participants Achieving Symptomatic Remission at Weeks 2, 4 and 8
Description: as for outcome 3
Time Frame: Weeks 2, 4 and 8
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Etrasimod 2 mg | Placebo
Number analyzed (Participants) | 222 | 112
Percentage of participants
  Week 2 | 16.2 | 10.7
  Week 4 | 27.5 | 16.1
  Week 8 | 38.7 | 24.1
Statistical Analysis 1: Comparison: Etrasimod 2 mg vs Placebo; Week 2; Test type: Superiority; p = 0.115, Cochran-Mantel-Haenszel; Risk Difference (RD) = 5.85, 95% CI 2-sided [-1.42 to 13.13]
Statistical Analysis 2: Comparison: Etrasimod 2 mg vs Placebo; Week 4; Test type: Superiority; p = 0.007, Cochran-Mantel-Haenszel; Risk Difference (RD) = 11.83, 95% CI 2-sided [3.19 to 20.47]
Statistical Analysis 3: Comparison: Etrasimod 2 mg vs Placebo; Week 8; Test type: Superiority; p = 0.003, Cochran-Mantel-Haenszel; Risk Difference (RD) = 14.84, 95% CI 2-sided [4.98 to 24.69]

8. Secondary Outcome: Percentage of Participants Achieving Complete Symptomatic Remission
Description: Complete symptomatic remission was defined as an SF sub-score = 0 and RB sub-score = 0. The SF sub-score ranged from 0 to 3 (where 0 = normal number of stools and 3 = at least 5 stools more than normal) and RB sub-score ranged from 0 to 3 (where 0 = no blood and 3 = blood alone passes). Higher scores indicated more severe disease.
Time Frame: Weeks 2, 4, 8 and 12
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Etrasimod 2 mg | Placebo
Number analyzed (Participants) | 222 | 112
Percentage of participants
  Week 2 | 4.5 | 1.8
  Week 4 | 11.7 | 3.6
  Week 8 | 14.0 | 7.1
  Week 12 | 18.0 | 8.9
Statistical Analysis 1: Comparison: Etrasimod 2 mg vs Placebo; Week 2; Test type: Superiority; p = 0.128, Cochran-Mantel-Haenszel; Risk Difference (RD) = 2.83, 95% CI 2-sided [-0.81 to 6.48]
Statistical Analysis 2: Comparison: Etrasimod 2 mg vs Placebo; Week 4; Test type: Superiority; p = 0.002, Cochran-Mantel-Haenszel; Risk Difference (RD) = 8.32, 95% CI 2-sided [3.01 to 13.64]
Statistical Analysis 3: Comparison: Etrasimod 2 mg vs Placebo; Week 8; Test type: Superiority; p = 0.032, Cochran-Mantel-Haenszel; Risk Difference (RD) = 7.06, 95% CI 2-sided [0.62 to 13.49]
Statistical Analysis 4: Comparison: Etrasimod 2 mg vs Placebo; Week 12; Test type: Superiority; p = 0.014, Cochran-Mantel-Haenszel; Risk Difference (RD) = 9.18, 95% CI 2-sided [1.82 to 16.54]

9. Secondary Outcome: Percentage of Participants Achieving Non-invasive Clinical Response
Description: Non-invasive clinical response was defined as a >= 30% decrease from Baseline in composite RB and SF sub-scores, and a >= 1 point decrease from Baseline in RB sub-score or RB sub-score <= 1. The SF subscore ranged from 0 to 3 (where 0 = normal number of stools and 3 = at least 5 stools more than normal) and RB sub-score ranged from 0 to 3 (where 0 = no blood and 3 = blood alone passes). The composite RB and SF score range was from 0 to 6, with higher scores indicating more severe disease.
Time Frame: Weeks 2, 4, 8 and 12
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Etrasimod 2 mg | Placebo
Number analyzed (Participants) | 222 | 112
Percentage of participants
  Week 2 | 39.2 | 24.1
  Week 4 | 55.9 | 41.1
  Week 8 | 68.0 | 45.5
  Week 12 | 67.6 | 50.0
Statistical Analysis 1: Comparison: Etrasimod 2 mg vs Placebo; Week 2; Test type: Superiority; p = 0.002, Cochran-Mantel-Haenszel; Risk Difference (RD) = 15.55, 95% CI 2-sided [5.65 to 25.46]
Statistical Analysis 2: Comparison: Etrasimod 2 mg vs Placebo; Week 4; Test type: Superiority; p = 0.007, Cochran-Mantel-Haenszel; Risk Difference (RD) = 14.98, 95% CI 2-sided [4.05 to 25.91]
Statistical Analysis 3: Comparison: Etrasimod 2 mg vs Placebo; Week 8; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Risk Difference (RD) = 22.60, 95% CI 2-sided [11.95 to 33.25]
Statistical Analysis 4: Comparison: Etrasimod 2 mg vs Placebo; Week 12; Test type: Superiority; p = 0.002, Cochran-Mantel-Haenszel; Risk Difference (RD) = 17.58, 95% CI 2-sided [6.70 to 28.47]

10. Secondary Outcome: Percentage of Participants Achieving Symptomatic Response
Description: Symptomatic response was defined as a >= 30% decrease from Baseline in composite RB and SF score. The SF sub-score ranged from 0 to 3 (where 0= normal number of stools and 3= at least 5 stools more than normal) and RB sub-score ranged from 0 to 3 (where 0= no blood and 3= blood alone passes). The composite RB and SF score range was from 0 to 6, with higher scores indicating more severe disease.
Time Frame: Weeks 2, 4, 8 and 12
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Etrasimod 2 mg | Placebo
Number analyzed (Participants) | 222 | 112
Percentage of participants
  Week 2 | 39.6 | 24.1
  Week 4 | 56.3 | 41.1
  Week 8 | 68.5 | 46.4
  Week 12 | 68.5 | 50.0
Statistical Analysis 1: Comparison: Etrasimod 2 mg vs Placebo; Week 2; Test type: Superiority; p = 0.002, Cochran-Mantel-Haenszel; Risk Difference (RD) = 15.99, 95% CI 2-sided [6.07 to 25.91]
Statistical Analysis 2: Comparison: Etrasimod 2 mg vs Placebo; Week 4; Test type: Superiority; p = 0.006, Cochran-Mantel-Haenszel; Risk Difference (RD) = 15.45, 95% CI 2-sided [4.54 to 26.36]
Statistical Analysis 3: Comparison: Etrasimod 2 mg vs Placebo; Week 8; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Risk Difference (RD) = 22.14, 95% CI 2-sided [11.43 to 32.85]
Statistical Analysis 4: Comparison: Etrasimod 2 mg vs Placebo; Week 12; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Risk Difference (RD) = 18.49, 95% CI 2-sided [7.65 to 29.33]

ADVERSE EVENTS:
Time Frame: All-cause mortality, non-serious Treatment-emergent adverse events (TEAEs) and Serious adverse events (SAEs) were collected from first dose of study intervention (Day 1) up to 30 days following discontinuation of the study intervention.
Description: Safety set population included all randomized participants who received at least 1 dose of study intervention.
Arm/Group | Etrasimod 2 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/238 | 0/116
Serious Adverse Events (participants affected / at risk) | 6/238 | 2/116
Other Adverse Events (participants affected / at risk) | 112/238 | 54/116
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Etrasimod 2 mg (N=238) | Placebo (N=116)
Colitis ulcerative (Gastrointestinal disorders) | 3 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Coronary artery disease (Cardiac disorders) | 1 | 0
Hepatobiliary procedural complication (Injury, poisoning and procedural complications) | 1 | 0
Migraine (Nervous system disorders) | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Etrasimod 2 mg (N=238) | Placebo (N=116)
Nausea (Gastrointestinal disorders) | 10 | 2
Colitis ulcerative (Gastrointestinal disorders) | 8 | 1
Vomiting (Gastrointestinal disorders) | 5 | 2
Abdominal pain (Gastrointestinal disorders) | 3 | 3
Diarrhoea (Gastrointestinal disorders) | 3 | 0
Flatulence (Gastrointestinal disorders) | 2 | 1
Abdominal tenderness (Gastrointestinal disorders) | 2 | 0
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1
Anal eczema (Gastrointestinal disorders) | 1 | 0
Frequent bowel movements (Gastrointestinal disorders) | 1 | 0
Gingival bleeding (Gastrointestinal disorders) | 1 | 0
Irritable bowel syndrome (Gastrointestinal disorders) | 1 | 0
Toothache (Gastrointestinal disorders) | 1 | 2
Chronic gastritis (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 1
Gastrointestinal hypermotility (Gastrointestinal disorders) | 0 | 1
Gastrointestinal pain (Gastrointestinal disorders) | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 1
Hyperaesthesia teeth (Gastrointestinal disorders) | 0 | 1
Lip blister (Gastrointestinal disorders) | 0 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 1
Urinary tract infection (Infections and infestations) | 4 | 0
COVID-19 (Infections and infestations) | 3 | 3
Upper respiratory tract infection (Infections and infestations) | 2 | 1
Sinusitis (Infections and infestations) | 2 | 0
Nasopharyngitis (Infections and infestations) | 3 | 2
Anal abscess (Infections and infestations) | 1 | 0
Campylobacter infection (Infections and infestations) | 1 | 0
Clostridium difficile colitis (Infections and infestations) | 1 | 0
Clostridium difficile infection (Infections and infestations) | 1 | 0
Cytomegalovirus infection (Infections and infestations) | 1 | 0
Cystitis (Infections and infestations) | 1 | 0
Conjunctivitis (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0
Genitourinary tract infection (Infections and infestations) | 1 | 0
Hordeolum (Infections and infestations) | 1 | 0
Infected dermal cyst (Infections and infestations) | 1 | 1
Influenza (Infections and infestations) | 1 | 0
Localised infection (Infections and infestations) | 1 | 0
Rhinitis (Infections and infestations) | 1 | 0
Oral herpes (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 0 | 2
Enterocolitis bacterial (Infections and infestations) | 0 | 1
Laryngitis (Infections and infestations) | 0 | 1
Rash pustular (Infections and infestations) | 0 | 1
Tooth infection (Infections and infestations) | 0 | 1
Viral infection (Infections and infestations) | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 5 | 0
Alanine aminotransferase increased (Investigations) | 3 | 0
Blood creatine phosphokinase increased (Investigations) | 3 | 1
Blood alkaline phosphatase increased (Investigations) | 2 | 0
Aspartate aminotransferase increased (Investigations) | 2 | 0
Activated partial thromboplastin time prolonged (Investigations) | 2 | 0
Blood bilirubin increased (Investigations) | 2 | 0
Blood cholesterol increased (Investigations) | 2 | 1
Blood triglycerides increased (Investigations) | 2 | 0
Weight decreased (Investigations) | 2 | 0
Blood glucose increased (Investigations) | 1 | 0
Blood pressure increased (Investigations) | 1 | 0
Blood thyroid stimulating hormone increased (Investigations) | 1 | 0
Blood thyroid stimulating hormone decreased (Investigations) | 1 | 1
Heart rate increased (Investigations) | 1 | 0
Heart rate decreased (Investigations) | 1 | 0
Hepatic enzyme increased (Investigations) | 1 | 0
Prothrombin time prolonged (Investigations) | 1 | 0
Liver function test abnormal (Investigations) | 1 | 0
International normalised ratio increased (Investigations) | 1 | 0
Pulmonary function test decreased (Investigations) | 1 | 0
Transaminases increased (Investigations) | 1 | 0
Blood creatinine increased (Investigations) | 0 | 1
FEV1/FVC ratio decreased (Investigations) | 0 | 1
Lipase increased (Investigations) | 0 | 1
Lung diffusion test decreased (Investigations) | 0 | 2
Headache (Nervous system disorders) | 11 | 2
Platelet count increased (Investigations) | 0 | 1
Somnolence (Nervous system disorders) | 3 | 1
Dizziness (Nervous system disorders) | 3 | 0
Dizziness postural (Nervous system disorders) | 1 | 0
Drug withdrawal headache (Nervous system disorders) | 1 | 0
Migraine (Nervous system disorders) | 1 | 4
Sinus headache (Nervous system disorders) | 1 | 0
Presyncope (Nervous system disorders) | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 14 | 8
Iron deficiency anaemia (Blood and lymphatic system disorders) | 3 | 3
Blood loss anaemia (Blood and lymphatic system disorders) | 1 | 0
Microcytic anaemia (Blood and lymphatic system disorders) | 1 | 0
Thrombocytosis (Blood and lymphatic system disorders) | 1 | 0
Fatigue (General disorders) | 3 | 0
Pyrexia (General disorders) | 8 | 3
Chest discomfort (General disorders) | 1 | 1
Feeling abnormal (General disorders) | 1 | 0
Injection site reaction (General disorders) | 1 | 0
Malaise (General disorders) | 1 | 1
Non-cardiac chest pain (General disorders) | 1 | 1
Thirst (General disorders) | 1 | 0
Asthenia (General disorders) | 0 | 1
Vaccination site pain (General disorders) | 0 | 1
Oedema peripheral (General disorders) | 0 | 1
Oedema (General disorders) | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 2 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 3
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 4 | 0
Iron deficiency (Metabolism and nutrition disorders) | 3 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 2 | 0
Folate deficiency (Metabolism and nutrition disorders) | 1 | 0
Gout (Metabolism and nutrition disorders) | 1 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Hypoproteinaemia (Metabolism and nutrition disorders) | 1 | 0
Hypovolaemia (Metabolism and nutrition disorders) | 1 | 0
Underweight (Metabolism and nutrition disorders) | 1 | 0
Increased appetite (Metabolism and nutrition disorders) | 1 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1
Uveitis (Eye disorders) | 2 | 0
Vision blurred (Eye disorders) | 2 | 0
Blepharitis (Eye disorders) | 1 | 0
Conjunctival haemorrhage (Eye disorders) | 1 | 0
Eye pain (Eye disorders) | 1 | 0
Conjunctivitis allergic (Eye disorders) | 1 | 0
Eyelid margin crusting (Eye disorders) | 1 | 0
Glaucoma (Eye disorders) | 1 | 1
Meibomian gland dysfunction (Eye disorders) | 1 | 0
Macular oedema (Eye disorders) | 1 | 1
Macular hole (Eye disorders) | 1 | 0
Visual impairment (Eye disorders) | 1 | 0
Pigment dispersion syndrome (Eye disorders) | 1 | 0
Metamorphopsia (Eye disorders) | 1 | 0
Visual snow syndrome (Eye disorders) | 1 | 0
Chorioretinopathy (Eye disorders) | 0 | 1
Exudative retinopathy (Eye disorders) | 0 | 1
Ocular hypertension (Eye disorders) | 0 | 1
Sinus bradycardia (Cardiac disorders) | 4 | 0
Tachycardia (Cardiac disorders) | 2 | 2
Atrioventricular block first degree (Cardiac disorders) | 1 | 0
Bradycardia (Cardiac disorders) | 1 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 0
Sinus arrhythmia (Cardiac disorders) | 1 | 0
Palpitations (Cardiac disorders) | 1 | 1
Ventricular extrasystoles (Cardiac disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0
Cutaneous vasculitis (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 0
Nail bed bleeding (Skin and subcutaneous tissue disorders) | 1 | 0
Miliaria (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0
Liver disorder (Hepatobiliary disorders) | 3 | 0
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 | 1
Blister (Skin and subcutaneous tissue disorders) | 0 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 0
Hepatic cytolysis (Hepatobiliary disorders) | 1 | 0
Cholestasis (Hepatobiliary disorders) | 1 | 0
Hypertension (Vascular disorders) | 3 | 1
Venous thrombosis (Vascular disorders) | 1 | 0
Essential hypertension (Vascular disorders) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 0
Vaccination complication (Injury, poisoning and procedural complications) | 1 | 1
Wound complication (Injury, poisoning and procedural complications) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Ear pain (Ear and labyrinth disorders) | 1 | 0
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 1 | 0
Testicular torsion (Reproductive system and breast disorders) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 | 0
Hyperthyroidism (Endocrine disorders) | 1 | 0
Food allergy (Immune system disorders) | 1 | 0
Papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Initial insomnia (Psychiatric disorders) | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 5 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-02-22): https://cdn.clinicaltrials.gov/large-docs/69/NCT03996369/Prot_000.pdf
  • Statistical Analysis Plan (2022-01-19): https://cdn.clinicaltrials.gov/large-docs/69/NCT03996369/SAP_001.pdf